CLINICAL TRIAL: NCT03323086
Title: Reducing Alcohol-related HIV/STI Risk for Women in Reproductive Health Clinics
Brief Title: Women SHARE Study: Reducing Sexual Risk
Acronym: HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Planned Parenthood of Southern New England (Other); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Michael P. Carey, Professor and Director, Centers for Behavioral and Preventive Medicine, The Miriam Hospital, The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 775844-4; R34AA023158 (NIH)
Record Dates: First submitted 2017-10-18; First posted 2017-10-26 (Actual); Results first posted 2020-01-02 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Alcohol and Substance-Related Mental Disorders; Sexually Transmitted Diseases
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention (BI) with Technology Extender (Experimental): Participants assigned to BI condition will receive a face to face session lasting 45-60 minutes delivered by a health coach. Following the session, participants will be given access to a study website and receive texts-of-the day on study topics.
  Interventions: Behavioral: Brief Intervention (BI) with Technology Extender
- Brochure (Other): Participants assigned to the Brochure condition will receive materials prepared by the Centers for Disease Control and Prevention on the study topics.
  Interventions: Other: Brochure

INTERVENTIONS:
Behavioral: Brief Intervention (BI) with Technology Extender — One, 45-60 minute BI, followed by three months of access to technology extenders
  Arms: Brief Intervention (BI) with Technology Extender
Other: Brochure — Brochures provided one time
  Arms: Brochure

SUMMARY:
This study will investigate whether BI and technology extenders are feasible and acceptable for female patients at a reproductive health center (ages 18-29).

DETAILED DESCRIPTION:
This study will assess the feasibility and acceptability, and obtain initial evidence of the efficacy, of the BI and technology extenders. At-risk women drinkers (N = 50) recruited from a reproductive health care clinic will be assessed, randomly assigned to the integrated BI or control (a Centers for Disease Control and Prevention-produced brochure with information about alcohol and women's health), and reassessed at 3 months to determine impact on alcohol use, condom use, and number of partners as well as hypothesized mediators.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age 18-29 years
* Meeting NIAAA definition of "at-risk" drinking (>3 drinks on any day in the last 3 months18 and/or >7 drinks per week)
* Sexual risk behavior (i.e., last 3 months: vaginal/anal intercourse with >1 partner; vaginal/anal intercourse with a partner who has other partners; inconsistent condom use; new relationship (under 3 months))
* English speaking
* Absence of acute intoxication, depression, or suicidal ideation
* No plans for relocation

Exclusion Criteria:

* Male
* Under 18 years old or older than 29 years old
* Non-English speaking
* Suicidal Ideation
* Relocating
* Clinic provider advising against recruitment in the study
* Unwilling or unable to provide consent

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — sex assigned at birth
Enrollment: 50 (Actual)
Dates: Start 2017-10-18 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Carey, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Planned Parenthood of Southern New England, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 women enrolled in the trial. Two women who enrolled withdrew prior to randomization. Thus, 48 women were randomized.
Period: Overall Study
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Started | 26 | 22
Completed | 23 | 20
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.28 (2.61) | 24.33 (2.92) | 22.67 (3.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 14
  Not Hispanic or Latino | 17 | 15 | 32
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 16 | 12 | 28
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Providing Intervention
Description: percentage of individuals who attended their intervention
Time Frame: Immediately following intervention session (post-intervention), up to 30 minutes
Population: 50 patients enrolled. 2 patients withdrew prior to randomization. Leaving 48 participants for this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Number analyzed (Participants) | 26 | 22
Participants | 25 | 22

2. Secondary Outcome: Session Evaluation Questionnaire
Description: Measure Name: Session Evaluation Questionnaire; Construct Assessed: Treatment Satisfaction; Minimum total scale score = 1; Maximum total scale score = 5; Scoring: averaged ratings across 4 items; Interpretation: Higher scores represent a better outcome.
Time Frame: Immediately following intervention session (post-intervention), up to 30 minutes
Population: 50 patients enrolled. However, 2 patients withdrew prior to randomization and 2 withdrew post-randomization leaving a total of 46 patients who provided data at this post-intervention assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Number analyzed (Participants) | 25 | 21
units on a scale | 4.65 (0.36) | 3.98 (0.96)

3. Secondary Outcome: Number of Sexual Partners
Description: The number of male partners that the participant reported having penetrative sex with.
Time Frame: 3-month Follow-up
Population: 50 patients enrolled. However, 2 patients withdrew prior to randomization, 2 withdrew post-randomization, and 3 were lost to follow-up, leaving a total of 43 patients who provided data at this 3-month follow-up assessment.
Measure: Mean (Standard Deviation); unit: partners
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Number analyzed (Participants) | 23 | 20
partners | 3.23 (3.22) | 4.00 (3.08)

4. Secondary Outcome: Condomless Sex
Description: The number of occasions of condomless sex
Time Frame: 3-month Follow-up
Population: as for outcome 3
Measure: Median (99% Confidence Interval); unit: events of condomless sex
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Number analyzed (Participants) | 23 | 20
events of condomless sex | 3 [2 to 4] | 5 [4 to 6]

5. Secondary Outcome: Alcohol Use Quantity
Description: The average number of drinks in a week
Time Frame: 3-month Follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: drinks per week
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Number analyzed (Participants) | 23 | 20
drinks per week | 3.23 (3.22) | 4.00 (3.08)

6. Secondary Outcome: Alcohol Use Binge Frequency
Description: The number of drinking occasions (single day) when 4 or more drinks are consumed
Time Frame: 3-month Follow-up
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: heavy episodic drinking days
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
Number analyzed (Participants) | 23 | 20
heavy episodic drinking days | 2.36 (3.27) | 2.00 (2.00)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Brief Intervention (BI) With Technology Extender | Brochure
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 0/26 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03323086/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-28): https://cdn.clinicaltrials.gov/large-docs/86/NCT03323086/SAP_001.pdf
  • Informed Consent Form (2017-10-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT03323086/ICF_002.pdf